CLINICAL TRIAL: NCT06509906
Title: An Open Label, Multicenter, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetic/Pharmacodynamic Profile of the PARP1 Inhibitor M9466 in Combination With Topoisomerase 1 Inhibitor-based Regimens in Advanced Solid Tumors and Colorectal Cancer (DDRiver 511)
Brief Title: M9466 in Combination With Topoisomerase 1 Inhibitors-based Regimens in Advanced Solid Tumors and Colorectal Cancer (DDRiver 511)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS202650_0001; 2024-514155-15-00 (Other: EU CTR)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumor
Keywords: PARP inhibitor; DNA repair inhibitor; Irinotecan; FOLFIRI
MeSH Terms: interventions — Irinotecan; Leucovorin; Fluorouracil; Bevacizumab; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- M9466 + Irinotecan (Run-in Cohort) (Experimental)
  Interventions: Drug: M9466; Drug: Irinotecan; Drug: Granulocyte colony stimulating factor (G-CSF)
- M9466 + FOLFIRI (folinic acid, fluorouracil, irinotecan) + Bevacizumab (Dose Finding Cohorts) (Experimental)
  Interventions: Drug: M9466; Drug: Irinotecan; Drug: Folinic acid; Drug: Fluorouracil (5-FU); Drug: Bevacizumab; Drug: Granulocyte colony stimulating factor (G-CSF)

INTERVENTIONS:
Drug: M9466 — M9466 will be administered orally until progressive disease, unacceptable toxicity, death, or end of study.
  Other Names: HRS-1167
Drug: Irinotecan — Irinotecan will be administered intravenously once every 2 weeks (q2w) until progressive disease, unacceptable toxicity, death, or end of study.
Drug: Folinic acid — Folinic acid will be administered intravenously q2w as per standard of care.
  Other Names: Calcium folinate Leucovorin
  Arms: M9466 + FOLFIRI (folinic acid, fluorouracil, irinotecan) + Bevacizumab (Dose Finding Cohorts)
Drug: Fluorouracil (5-FU) — Fluorouracil will be administered intravenously as per standard of care.
  Other Names: 5-FU
  Arms: M9466 + FOLFIRI (folinic acid, fluorouracil, irinotecan) + Bevacizumab (Dose Finding Cohorts)
Drug: Bevacizumab — Bevacizumab will be administered intravenously, q2w until progressive disease, unacceptable toxicity, death, or end of study.
  Arms: M9466 + FOLFIRI (folinic acid, fluorouracil, irinotecan) + Bevacizumab (Dose Finding Cohorts)
Drug: Granulocyte colony stimulating factor (G-CSF) — G-CSF will be administered subcutaneously at every cycle of study intervention as per standard of care.

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary clinical activity of M9466 in combination with topoisomerase 1 inhibitors-based regimens. As such the combination with FOLFIRI (folinic acid, fluorouracil, irinotecan) and Bevacizumab will be evaluated in participants with colorectal cancer, to establish the M9466 maximum tolerated dose if observed and the recommended dose for expansion.

Study Duration: After a Screening period of up to 28 days, enrolled participants will remain in the study until they have completed all the study visits or until they withdraw consent, are lost to follow-up, or die.

Visit Frequency: The participants will come for a Screening Visit and 1 to 2 visits per treatment cycle. After end of study intervention period, the participants will come for an End of Treatment Visit and a Safety Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* M9466 + Irinotecan Run-in Cohort: Participants with locally advanced or metastatic disease that is refractory to standard therapy or for which no standard therapy is judged appropriate by the Investigator (that is [i.e.] participants who have exhausted all standard of care (SoC) options according to International Guidelines), and who may derive clinical benefit from the combination treatment with M9466 and irinotecan
* M9466 + FOLFIRI + Bevacizumab Dose Finding Cohorts: Participants with documented histopathological diagnosis of locally advanced or metastatic colorectal cancer (CRC), who were intolerant/refractory to or progressed after standard systemic therapies for the advanced/metastatic stage that included: Oxaliplatin and a fluoropyrimidine (administration in the adjuvant setting fulfills this criterion if progression occurred within 12 months of the last dose). Prior use of irinotecan is permitted; Either an anti- epidermal growth factor receptor (anti-EGFR) or an anti- Vascular endothelial growth factor (anti-VEGF) agent (not applicable if oxaliplatin was administered in the adjuvant setting); An immune checkpoint inhibitor for participants with known MSI-H status; Anti-EGFR agent and BRAF tyrosine kinase inhibitor ± MEK inhibitor, if locally available, for participants with BRAF V600E mutations. Participants may have received maximally 1 previous regimen for the treatment of metastatic disease (with the exception of participants with MSI-H disease or BRAF positive disease who are allowed to have had up to 2 previous lines of treatment)
* Eastern Cooperative Oncology Group performance status (ECOG PS) less than or equal to (<=) 1
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Persistence of AEs related to any prior treatments that have not recovered to Grade <= 1 by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) unless AEs are clinically nonsignificant and/or stable on supportive therapy in the opinion of the Investigator (for example [e.g.] neuropathy or alopecia)
* History of additional malignancy within 3 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, benign prostate neoplasm/hypertrophy, or malignancy that in the opinion of the Investigator, is considered cured with minimal risk of recurrence within 3 years). Participants with history of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) are excluded, irrespective of timeframe
* Participant with known polymorphisms in UGT1A1, DPYD or other enzymes known to predict for increased toxicity from irinotecan or 5 fluorouracil (5-FU) should be excluded; if status is unknown testing is not mandated, unless required by local guidance. Participants that discontinued prior 5-FU treatment due to toxicity are also excluded
* Participants with known brain metastases, except if clinically controlled, which is defined as individuals with central nervous system (CNS) tumors that have been treated and are asymptomatic, and who have discontinued steroids (for the treatment of CNS tumors) for > 28 days prior to first dose of study intervention
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Treatment Related TEAEs | Time from signing Informed Consent Form (ICF) up to 30 days after end of study intervention (approximately assessed up to 18.7 months)
Number of Participants with Dose Limiting Toxicity (DLT) | Day 1 up to Day 28 of the first two Cycles (each cycle is of 14 days)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Plasma Concentration of M9466 | Pre-dose up to 6 hours post-dose on Cycle 1 Day 1; (each cycle is of 14 days)
Objective Response (OR) According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) Assessed by Investigator | Time from first treatment of study intervention up to planned assessment at 18.7 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc.
Locations (12):
- United States (4):
  - Sarah Cannon Research Institute at Health One, Denver, Colorado
  - Carolina BioOncology Institute, LLC - Cancer Therapy and Research Center, Pennington, New Jersey
  - Vanderbilt University - 150912667, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Cancer Research SA, Elizabeth Vale
  - St George Private Hospital, Kogarah
  - Peter MacCallum Cancer Centre - Use the one with Account 2 VCCC, Parkville
- National Cancer Center Hospital, Chūōku, Japan
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (2):
  - NEXT Barcelona - NEXT Barcelona, Barcelona
  - NEXT Madrid - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202650_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html